CLINICAL TRIAL: NCT01189084
Title: An Observational Study to the Patients With Alzheimer's Disease Who Previously Received UB311-Treatment in the V118-AD Trial
Brief Title: Observational Study to Monitor Long-term Immunogenicity and Efficacy of UB 311 Vaccine in Subjects With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: United Biomedical (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); National Taiwan University Hospital (Other)
Responsible Party: Pei-Ning Wang, M.D., Principal Investigator, Taipei Veterans General Hospital (TVGH)
Other Study IDs: UBI Protocol V118-obs
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; amyloid beta; vaccine
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Periodic blood samples collected for serum and measurement of anti-Amyloid-beta antibody levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational immunotherapy follow-up
  Interventions: Biological: Observational

INTERVENTIONS:
Biological: Observational — Measure anti-Amyloid-beta antibody in serum during 24-26 weeks extension period to 48 weeks (after first vaccine treatment).

SUMMARY:
The purpose of this observational study is to determine whether the vaccine (UB 311), targeting the N-terminal amino acids (1-14) of the amyloid beta peptide, has long-term immunogenicity and efficacy in individuals diagnosed with mild or moderate Alzheimer's disease (AD) who previously received UB 311-treatment. Amyloid beta was selected as the target antigen based on supporting evidence of the hypothesis that places the accumulation of amyloid beta at the initiating step of AD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with mild to moderate Alzheimer's disease who received three (3) injections of UB 311 in the initial Phase I V118-AD trial

Exclusion Criteria:

* Individuals with Alzheimer's disease who are currently on prohibited medications, have severe or uncontrolled systemic disease, or are unable or unwilling to comply with study protocol requirements.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled subjects who received UB 311-treatment in the initial UBI Protocol V118 (Protocol V118-AD) Phase I trial are eligible for continued follow-up to week 48
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-04; Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 24 weeks
  Long-term followup to week 48

SECONDARY OUTCOMES:
Efficacy | 24 weeks
  Long-term followup to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ning Wang, M.D., Principal Investigator — Taipei Veterans General Hospital (TVGH); Ming-Jang Chiu, M.D., Principal Investigator — National Taiwan University Hospital (NTUH)
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital (NTUH), Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Background] Wang CY, Finstad CL, Walfield AM, Sia C, Sokoll KK, Chang TY, Fang XD, Hung CH, Hutter-Paier B, Windisch M. Site-specific UBITh amyloid-beta vaccine for immunotherapy of Alzheimer's disease. Vaccine. 2007 Apr 20;25(16):3041-52. doi: 10.1016/j.vaccine.2007.01.031. Epub 2007 Jan 19. PMID 17287052
- See also: ClinicalTrials.gov Identifier: NCT00965588 — http://ClinicalTrials.gov